CLINICAL TRIAL: NCT04542590
Title: A Natural History Study of Patients With Genetically Confirmed Primary Hyperoxaluria Type 3 and, as Applicable Per Age, a History of Stone Events
Brief Title: Natural History of Patients With PH3 and a History of Stone Events
Acronym: PHYOX-OBX
Status: Completed | Type: Observational
Sponsor: Dicerna Pharmaceuticals, Inc., a Novo Nordisk company (Industry)
Responsible Party: Sponsor
Organization: Novo Nordisk A/S (Industry)
Other Study IDs: DCR-PHXC-502
Record Dates: First submitted 2020-08-20; First posted 2020-09-09 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Primary Hyperoxaluria Type 3
Keywords: primary hyperoxaluria; PH3; observational; kidney stones; nephrocalcinosis
MeSH Terms: conditions — Hyperoxaluria, Primary; Kidney Calculi; Nephrocalcinosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a natural history study of adults, adolescents, and children (starting at birth) with genetically confirmed primary hyperoxaluria type 3 (PH3) who have a history of stone events during the last 3 years and/or the presence of pre existing stones detected by renal ultrasound at screening.

DETAILED DESCRIPTION:
The relationship between the level of Uox and the incidence of kidney stones and/or nephrocalcinosis in patients with PH3 has not been established. The goal of this study is to record 24-hour Uox levels and the incidence of new stone formation and/or the degree of nephrocalcinosis in patients with PH3 over time.

Potential participants are screened over an up-to-7 week period according to the eligibility criteria and will then be followed every 6 months over an up-to-2-year period to determine the annualized new stone formation rate (number of new stones being formed per year) and the change in the degree of nephrocalcinosis (if applicable).

New stone formation is defined as occurrence of any of the following:

* Spontaneous stone passage in the absence of pre-existing stones
* Stone passage occurring without change in the number of pre-existing stones detected by renal ultrasound
* Appearance of new stones on renal ultrasound or 100% or more growth of a pre-existing stone (estimated area)
* Surgical removal of newly formed stones Note: Spontaneous passage or surgical removal of pre-existing stones does not meet the criteria for new stone formation.

This is a non-interventional study that will last up to 2 years.

ELIGIBILITY:
Key inclusion criteria

* Genetically confirmed PH3
* For participants at least 2 years of age, history of stone events (defined as presence of calcifications in the urinary tract and/or kidney, their relative location, and the number and size of stones) during the last 3 years and/or presence of pre-existing stones detected by renal ultrasound at Screening
* Uox ≥ 0.7 mmol/24 hours (adjusted per 1.73 m2 BSA in participants < 18 years of age) OR if not able to collect 24-hour urine, average spot Uox to creatinine ratio at Screening above the 95th percentile for age:

  * > 220 mmol/mol in participants < 6 months
  * > 170 mmol/mol in participants from 6 months to < 12 months
  * > 130 mmol/mol in participants 12 months to < 2 years
  * > 100 mmol/mol in participants from 2 to < 3 years and
  * > 80 mmol/mol in participants from 3 to 5 years
* eGFR at Screening ≥ 30 mL/min or for infants aged less than 12 months, serum creatinine below the 97th percentile of a healthy population

Key Exclusion Criteria:

* Prior or planned liver transplant within study period
* Currently receiving dialysis or anticipating dialysis during study period
* Unwillingness to comply with study procedures

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This is a natural history study in adults, adolescents, and children (starting from birth) with genetically confirmed PH3 who have a history of stone events during the last 3 years and/or the presence of preexisting stones detected by renal ultrasounds at Screening, and an eGFR > 30 mL/min/1.73 m2 or serum creatinine below the 97th percentile for patients younger than 12 months old.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2024-07-23 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Collect stone formation data in PH3 patients | Assess participants' stone formation rates over the course of 2 years
  Collect data on the rate of new stone formation in PH3 patients of at least 2 years of age
Assess relationship between urine oxalate (Uox) levels and stone formations in PH3 patients | Measure participants' Uox levels over the course of 2 years
  Explore the potential relationship between Uox levels and new stone formation in patients (≥ 2 years of age) with genetically confirmed PH3 and relatively intact renal function
Collect data on the degree of nephrocalcinosis in PH3 patients | Assess the change in nephrocalcinosis grade over the course of 2 years
  Collect data on the degree of nephrocalcinosis in PH3 patients of at least 2 years of age

CONTACTS AND LOCATIONS:
Overall Officials: Verity Rawson, Study Director — Dicerna, A Novo Nordisk Company
Locations (6):
- United States (2):
  - Clinical Trial Site, Boston, Massachusetts
  - Clinical Trial Site, New York, New York
- Clinical Trial Site, Toronto, Ontario, Canada
- Clinical Trial Site, Heidelberg, Germany
- Clinical Trial Site, Warsaw, Poland
- Clinical Trial Site, London, United Kingdom